CLINICAL TRIAL: NCT03818568
Title: Restriction of Proteins in the Diet and Supplementation With Ketoanalogues to Prevent Disease Progression in Patients With Stage 4 Chronic Kidney Disease
Brief Title: Supplemented Low Protein Diet and Progression of CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Principal Investigator, Jose Ramon Paniagua Sierra, Chief investigator, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-785-038
Record Dates: First submitted 2018-06-07; First posted 2019-01-28 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Stage 4 Chronic Kidney Disease
Keywords: chronic kidney disease; ketoanalogue; diabetes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Design. A multicenter, controlled, randomized, open label clinical trial. Group were: Low Protein Diet (LPD) and LPD Supplemented with Ketoanalogs (LPD+KA). The follow-up period was 1 year.
  Inclusion criteria: Adult patients with Type 2 Diabetes Mellitus, either sex, in stage 3b-4 of CKD. Exclusion criteria: Previous treatment with KA, kidney transplantation, cancer, HIV-AIDS, hepatitis B or C, patients receiving immunosuppressors, hypercalcemia, intolerance to KA or disorders of amino acid metabolism.
  Intervention. In both groups diet composition was the same: Energy, 35 kcals/kg, Lipids 35% and, Carbohydrate 55-60% of the total energy intake, fiber 20-25 g, NaCl ~5 g, K 50-60, Phosphate 800-1000 mg. Protein intake was 0.6 g/kg/day.
  Patients in LPD+KA received KA (1 tablet/5 kg/day). Each tablet contains: Keto-analogs of Isoleucine, Leucine, Phenylalanine, and Valine; hydroxyl analog of Methionine, and aminoacids Lysine, Threonine, Tryptophan, Histidine, and Tyrosine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketoanalogues of essential amino acids (Experimental): Patients will receive conventional treatment according to the institution's clinical guidelines, with moderate restriction of proteins 0.6 g protein/kg/day, as recommended to slow renal damage progression), plus ketoanalogues in the established dosage (1 tablet/5 kg weight divided into 3 doses per day).
  Interventions: Dietary Supplement: ketoanalogues of essential amino acids
- Control (Active Comparator): Patients will receive conventional treatment according to the institution's clinical guidelines, with moderate restriction of proteins 0.6 g protein/kg/day, as recommended to slow renal damage progression).
  Interventions: Dietary Supplement: ketoanalogues of essential amino acids

INTERVENTIONS:
Dietary Supplement: ketoanalogues of essential amino acids — Patients will receive conventional treatment according to the institution's clinical guidelines, with moderate restriction of proteins 0.6 g protein/kg/day, as recommended to slow renal damage progression), plus ketoanalogues in the established dosage (1 tablet/5 kg weight divided into 3 doses per day).

SUMMARY:
Investigators intend to analyze diets restricted in protein and supplemented with ketoanalogues of essential amino acids, to slow the progress of renal damage and improve nutritional status in diabetic patients over 60 years with stage 4 chronic kidney disease.

Evey 2 months, evaluations were performed of renal function (creatinine clearance, serum cysteine, proteinuria) and nutritional status (subjective global evaluation,dominant had pressure strength, body composition by bioelectric impedance, serum transferrin, serum prealbumin and serum aminogram) for a follow-up period of 2 years.

DETAILED DESCRIPTION:
Design. A multicenter, controlled, randomized, open label clinical trial was performed in patients with T2DM in CKD stage 3b-4 (GFR <44 to >15 mL/min/1.73 m2) treated in hospitals of the Mexican Social Security Institute. The follow-up period was at least 1 year from the inclusion of the last patient. The study was conducted in accordance with the provisions of the Declarations of Helsinki and Tokyo with the amendments in Venice (1983). The protocol was approved by the National Research and Ethics Committee and by the Research Committees of all participating hospitals and was registered in National Clinical Trials (NCT03818568).

Patients. Inclusion criteria: Adult patients with T2DM (>18 years) of either sex, with stage 3b-4 of CKD. All patients gave their signed informed consent at the time of recruitment. Exclusion criteria: Previous treatment with KA, kidney transplantation, cancer, HIV-AIDS, or seropositive for hepatitis B or C, patients receiving immunosuppressors, with hypercalcemia, intolerance to KA or disorders of amino acid metabolism. Patients who lost social security during the study, changed address or treating physician were also excluded.

Sample size. Sample size calculation was made on the basis of two independent groups with unequal variances, α=0.05, β=0.20, and assuming a difference of 4.0 mL/min/yr between groups in reduction of eGFR, lower in LPD+KA. Calculation was made with sample size software. A minimum of 51 per group was obtained.

Intervention. Diet design. Energy: 35 kcals/kg of ideal body weight in patients with normal BMI; 30 kcals/kg of ideal body weight in overweight patients (BMI>25 kg/m2) and 40 kcals/kg of ideal weight in underweight patients (BMI<25 kg/m2). Lipids accounted for 35% of the total energy intake (2/3 from polyunsaturated fatty acids). Carbohydrate intake was set at 55-60% of the total energy intake, with >70% of complex carbohydrates. The fiber content was 20-25 g per day. The dietary recommendation for sodium chloride was ~5 g daily and potassium 50-60 mEq/day. Phosphate intake was set at 800-1000 mg per day.

Both groups were prescribed with PrI of 0.6 g/kg/day, preferably plant-based. Patients in LPD+KA group received KA (Ketosteril® (Fresenius Kabi, Deutschland GMBH, BadHomburg, Germany) according to the manufacturer's recommendations (1 tablet/5 kg of body weight divided into 3 doses). All other treatments were provided according to institutional guidelines and prescribed by and according to the criteria of the treating physicians.

Randomization. Patients were centrally randomized 1:1 using an electronic system of random numbers generator.

Outcomes. The primary outcome was: the rate of decline in kidney function (Δ eGFR/year). Secondary outcomes included: start of dialysis, impairment of nutritional status, adverse events, hospitalizations, and mortality.

Follow-up. Patients were followed-up with scheduled visits every two months, for clinical and biochemical evaluation. Blood samples were obtained after an overnight fast, serum and plasma were separated and kept in frozen aliquots (-70 °C) until assay. The 24 h urine volumes were recorded and frozen aliquots stored (-70 °C) until assay. In total blood, hemoglobin, hematocrit, and glycated hemoglobin were measured, and in plasma/serum: glucose, urea, creatinine, albumin, total proteins, triglycerides, total cholesterol, HDL cholesterol, calcium, phosphorus, C-reactive protein. In 24-hour urine: urea and creatinine. Serum Cystatin-C was measured at baseline and months 6, 9 and 12.

Measurements of biochemical parameters were performed on automated equipment using routine techniques. High sensitivity C-reactive protein and Cystatin-C were measured by immunoturbidimetry (Diazyme's Cystatin C Assay. Poway, CA, USA). The protein nitrogen appearance normalized by body weight (nPNA) was calculated with the Maroni formula, GFR was calculated using formulas based on sCr (eCKDCr), and serum Cystatin C (eGFRCysC).

Nutritional evaluations. The patients were evaluated by Nephrology Nutritionists. Nutritional status was monitored by body weight, body mass index, subjective global assessment, body composition analyzed by electrical bioimpedance, and biochemical parameters. As a functional index, the hand grip force was measured with a dynamometer. Treatment adherence was monitored by the 24-hour food intake questionnaire and/or the 3-day food intake diary, nPNA was also used. In the intervention group, adherence to the use of KA was evaluated by counting tablets and packaging at each visit.

Statistical analysis. Data are presented as means and standard deviations or standard errors and as percentages or frequencies according variable characteristics. Differences between groups were analyzed with Chi2 test, or Student´s t test. For calculation of decline of GFR during follow-up, only actual eGFR data were considered, and two-way analyses of variance used. For analysis of the effect of concomitant medication, differences in slopes of regression lines of eGFR over time among users and non-users of specific medication were used. Differences in distribution of adverse events was analyzed with Chi2 and Kolmogorov-Smirnov test. All statistical calculations were made with wSPSS v19 package.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetic nephropathy in stage 4 chronic kidney disease
* Patients in pre-dialysis
* Patients with signed informed consent forms.

Exclusion Criteria:

* Patients who have received Ketosteril previously
* Patients participating in other intervention studies
* Pregnant women
* Patients with background of renal transplant
* Patients with cancer, HIV, seropositive for hepatitis B or C or receiving immunosuppressors, hypercalcemia
* Intolerance of Ketosteril ingredients
* Hereditary disorders in amino acid metabolism

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
glomerular filtration | 2 years
  Speed of reduction in glomerular filtration measured by cysteine C clearance and the need for dialysis glomerular filtration <15 mL/min/1.73 m2)

SECONDARY OUTCOMES:
Comorbidities | 2 years
  measure of frequency and number of comorbidities
Hospitalizations | 2 years
  measure of number and length of hospitalizations
Mortality | 2 years
  measure of incidence of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Paniagua, MD, PhD, Study Director — Instituto Mexicano del Seguro Social
Locations (2):
- Mexico (2):
  - Unidad de Investigación Médica en Enfermedades Nefrológicas, Instituto Mexicano del Seguro Social, Mexico City, Mexico City
  - Unidad de Investigacion Medica en Enfermedades Nefrologicas, Hospital de Especialidades Centro Medico Nacional Siglo XXI, Mexico City

IPD SHARING:
Plan to Share IPD: No